CLINICAL TRIAL: NCT04188587
Title: 177Lu-PSMA-I＆T PSMA Radioligand Therapy in Metastatic Castration-Resistant Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, FengWang, Director of Nuclear Medicine, Nanjing First Hospital, Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: fengwang-177LU-PSMA
Record Dates: First submitted 2019-12-04; First posted 2019-12-06 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: 177Lu-PSMA-I&T; Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 177Lu-PSMA-I&T (Experimental): 177Lu-PSMA-I＆Tradioligand therapy with 2.0-8.0GBq in every circle were performed. And then 177Lu-PSMA post-therapy scans were performed at 24 h and 48 h respectively, and the fusion phenomenon was performed at the second day to pre evaluate the efficacy of the patients.
  Interventions: Drug: 177 Lu-PSMA-I&T

INTERVENTIONS:
Drug: 177 Lu-PSMA-I&T — All patients were intravenous injected with single dose 2.0-8.0 GBq. The time of the next treatment cycle is determined according to the patient's condition, and it is recommended to treat once every 8-12 weeks.

SUMMARY:
The purpose of this study is to determine the safety and efficacy of 177 Lu -labeled PSMA ligand(PSMA-I＆T) in the treatment of mCRPC in Asianethics.

DETAILED DESCRIPTION:
Prostate specific membrane antigen(PSMA) targeted therapy brings new hope to the patients with metastatic castration-resistant prostate cancer (mCRPC). Here, we reported the safety and efficacy of 177 Lu -labeled PSMA ligand(PSMA-I＆T) in the treatment of mCRPC in Asianethics.

Prostate cancer is the most common cancer diagnosed in older men with recent data .PSMA is a type II transmembrane glycoprotein，overexpressed up to 100 to 1000 times higher than normal prostate cells in prostate cancer cells and is correlated with higher-grade cancers, metastatic disease and hormone refractory disease. Lutetium-177 (177Lu)-PSMA (LuPSMA) is a novel and highly targeted systemic RLT for progressive mCRPC. Upon binding of LuPSMA to the cell membrane, endocytosis is triggered, concentrating the tumouricidal effects of the radioisotope activity internally within malignant cells.

This is a single-institution, single-arm phase 2 clinical trial. Patients will receive PRLT Treatment. The follow-up period was followed up to assess safety and effectiveness.

ELIGIBILITY:
Entry criteria

1. ECOG score: 0-1 point
2. Lymph and skeletal metastases or visceral metastases that cannot be removed surgically
3. The disease continues to progress after treatment with ADT, chemotherapy, radiotherapy, or abiraterone and emzaludine 4.68Ga PSMA-11 PET / CT showed that there was significant radioactivity uptake in tumor tissues and metastases [SUVmax> 7], which was significantly higher than that in the liver.

Exclusion criteria

1. Previous treatment with any of the following within 6 months of randomization:

   Strontium-89, Samarium-153, Rhenium-186, Rhenium-188, Radium-223, hemi-body irradiation. Previous PSMA-targeted radioligand therapy is not allowed.
2. Hemoglobin<80g/L;Hemameba<2.5×109/L;Thrombocyte<70g/L
3. Glomerular filtration rate<50ml/min
4. Serum creatinine>130umol/L;Total bilirubin>2mg/L;Albumin<30g/L.
5. International normalized ratio（INR）>1,5
6. Alanine aminotransferase, aspartate aminotransferase is 5 times larger than normal value

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
PSA | 2 months
  Serum prostate specific antigen (PSA) levels was used as the main marker of efficacy evaluation, and the changes of PSA level were divided into decrease > 50%, 30% ~ 50% and < 30%.

SECONDARY OUTCOMES:
Adverse events collection | 2 months
  Adverse events within 2 months after the injection and scanning of patients will be followed and assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China